CLINICAL TRIAL: NCT04675983
Title: A Randomized, Multicenter, Phase 3 Study to Evaluate the Efficacy and Safety of Sintilimab Combined With Ramucirumab as Compared to Chemotherapy for the First-line Treatment of Unresectable Locally Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma (ORIENT-106)
Brief Title: A Study of Sintilimab Plus Ramucirumab as First-line Treatment for G/EGJ Adenocarcinoma (ORIENT-106)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the company's development strategy adjustment, Innovent Biologics has decided not to continue this study after consultation with investigators
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI308E302
Record Dates: First submitted 2020-12-03; First posted 2020-12-19 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Gastric Adenocarcinoma
MeSH Terms: interventions — sintilimab; Ramucirumab; Cisplatin; Fluorouracil; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab + Ramucirumab (Experimental): Ramucirumab on days 1 and 8 in combination with Sintilimab on day 1 of each 21-day cycle until disease progression, intolerable toxicity or other criteria for treatment discontinuation
  Interventions: Drug: Sintilimab; Drug: Ramucirumab
- Cisplatin+ 5-fluorouracil/Oxaliplatin+capecitabine (Active Comparator): Cisplatin on day 1 in combination with 5-fluorouracil, continuous pumping for 24 hours a day on days 1 to 5 of each 21-day cycle. (FP regimen) or Oxaliplatin on day 1 in combination with capecitabine on days 1 to 14 of each 21-day cycle. (XELOX regimen)
  Interventions: Drug: Cisplatin; Drug: 5-fluorouracil; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Sintilimab — Administered IV
  Other Names: Tyvyt; IBI308
  Arms: Sintilimab + Ramucirumab
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806; IMC-1121B; Cyramza
  Arms: Sintilimab + Ramucirumab
Drug: Cisplatin — Administered IV
  Arms: Cisplatin+ 5-fluorouracil/Oxaliplatin+capecitabine
Drug: 5-fluorouracil — Administered IV
  Arms: Cisplatin+ 5-fluorouracil/Oxaliplatin+capecitabine
Drug: Oxaliplatin — Administered IV
  Arms: Cisplatin+ 5-fluorouracil/Oxaliplatin+capecitabine
Drug: Capecitabine — Administered orally
  Arms: Cisplatin+ 5-fluorouracil/Oxaliplatin+capecitabine

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of sintilimab plus ramucirumab compared to stand of care first-line chemotherapy in participants with advanced gastric or esophagogastric adenocarcinoma.

DETAILED DESCRIPTION:
This is a randomized, multicenter, phase 3 study to evaluate the efficacy and safety of sintilimab combined with ramucirumab as compared to stand of care chemotherapy for the first-line treatment of PD-L1 positive, unresectable locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma.

The primary endpoint of this study is OS of the ITT population.

ELIGIBILITY:
Inclusion criteria

* Have a histologically confirmed diagnosis of gastric or gastroesophageal junction adenocarcinoma
* With HER2 negative and PD-L1 positive tumor tissue
* Have fresh or archival tumor tissue samples within 6 months for PD-L1 expression test.
* Age ≥18 and ≤75 years
* Diagnosed as unresectable locally advanced or metastatic stage

Exclusion criteria

* Have received any prior palliative systemic treatment for advanced gastric or gastroesophageal junction adenocarcinoma.
* Known to have central nervous system metastases, cancerous meningitis, or bone metastases with a risk of paraplegia
* Known bone metastasis with a risk of paraplegia.
* Have any ascites that requires intervention.
* With bilateral medium pleural effusion or unilateral large pleural effusion leading to respiratory symptoms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-02-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of sintilimab plus ramucirumab,Overall survival (OS) | Randomization to Death from Any Cause, up to 60 months
  OS is time from the date of randomization to the date of death from any cause. If the participant is alive at the cutoff for analysis (or was lost to follow-up), OS data is censored for analysis on the last date the participant is known to be alive.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Randomization to Radiological Disease Progression or Death from Any Cause (Up to 24 Months)
  PFS is time from the date of randomization to the date of radiographic documentation of progression (per RECIST v.1.1) or the date of death due to any cause, whichever is earlier. If a participant is not known to have died or have radiographic documented progression as of the data cutoff date for the analysis, the PFS time is censored at the last adequate tumor assessment date.
Objective Response Rate [ORR] (Percentage of Participants With Complete Response [CR] or Partial Response [PR]) | Randomization to Disease Progression (Up To 24 Months)
  Response is defined using RECIST v1.1. ORR is calculated as sum of the number of participants with CR and PR divided by the number of evaluable participants multiplied by 100.
Disease Control Rate [DCR] (Percentage of Participants With Complete Response [CR], Partial Response [PR] or Stable Disease [SD]) | Randomization to Disease Progression (Up To 24 Months)
  Response is defined using RECIST v1.1. DCR is calculated as sum of the number of participants with CR, PR, and SD divided by the number of evaluable participants multiplied by 100.
Duration of Response (DoR) | Date of Complete Response (CR) or Partial Response (PR) to Date of Objective Disease Progression or Death Due to Any Cause (Up To 24 Months)
  DoR is time from the date of first radiographic documentation of CR or PR to the date of first radiographic documentation of PD or death due to any cause. If a participant is not known to have died or have radiographically documented PD as of the data inclusion cutoff date, DOR is censored at the date of the last adequate tumor assessment.
Number of participants experiencing an adverse event (AE) | Randomization to end of study (up to 24 months)
  An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. The number of participants who experienced an AE is reported for each arm according to the treatment received.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China